CLINICAL TRIAL: NCT03473496
Title: The Prospective, Multi-center And Single-arm Clinical Study of Chimeric Antigen Receptor T(CAR-T) Cells Therapy in Relapsed/Refractory Multiple Myeloma
Brief Title: CAR-T Cells Therapy in Relapsed/Refractory Multiple Myeloma
Acronym: MM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: After CAR-T treatment, the benefit is not significant, and it is difficult to enroll.
Sponsor: Zhujiang Hospital (Other)
Collaborators: Nanfang Hospital, Southern Medical University (Other); The Third Affiliated Hospital of Southern Medical University (Other Government); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-XYNK-003
Record Dates: First submitted 2018-03-15; First posted 2018-03-22 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2021-09

CONDITIONS: Relapsed/Refractory Multiple Myeloma(MM)
Keywords: BCMA-CART; CD138-CART; CD56-CART; CD38-CART
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CART therapy in multiple myeloma (Experimental): In order to assess the safety and validity of using CAR-T therapy refractory/rela-psed multiple myeloma patients with one kind of BCMA-CART,CD138-CART,CD56-CART or CD38-CART,subjects will receive 10^6-10^7/Kg transduced CAR T cells at one time.
  Interventions: Biological: CART therapy in Relapsed/Refractory multiple myeloma

INTERVENTIONS:
Biological: CART therapy in Relapsed/Refractory multiple myeloma — one kind of BCMA/CD138/CD38/CD56-CART therapy in Relapsed/Refractory multiple myeloma

SUMMARY:
Multiple myeloma（MM） is one of the most common malignant diseases in the blood system.There is still no cure for the disease which only control the development of the disease in various ways.Chimeric Antigen Receptor-transduced T cell (CAR-T) therapy is one of revolutionary targeted immunotherapy.The efficacy of CAR-T cells for the treatment of acute B lymphocytic leukemia has been widely recognized, and several clinical trials have been reported in the treatment of multiple myeloma with CAR-T cells.

DETAILED DESCRIPTION:
Multiple myeloma（MM） is one of the most common malignant diseases in the blood system.There is still no cure for the disease which only control the development of the disease in various ways.

In recent years, the understanding of pathogenic molecular mechanism in MM , many new types of drugs can be used in the treatment of this disease, one of the most widely used is proteasome inhibitors and immune regulator.Hematopoietic stem cell transplantation has also been shown to improve complete remission rates and prolong patient survival.Combined with the advantages of multiple therapies, chimeric antigen receptor T cells (CAR-T) have gradually become one of the strongest and most powerful weapons against multiple myeloma.

CAR - T cells was taken in the form of genetic modification, and specific identified target antigen monoclonal antibody of single variable region (scFv) expression in T cell surface, and coupled with the activation of intracellular proliferation signal domain.

When scFv recognizes antigens expressed in malignant cells, it stimulates the activation signal of downstream T cells and produces specific killing effects. CAR-T therapy is one of revolutionary targeted immunotherapy.The efficacy of CAR-T cells for the treatment of acute B lymphocytic leukemia has been widely recognized, and several clinical trials have been reported in the treatment of multiple myeloma with CAR-T cells.Throughout registration of clinical trials and published research results, B-cell maturation antigen (BCMA) as one of targets , its effect is more significant than other molecules.As with BCMA antigens, cluster of differentiation 138(CD138), cluster of differentiation 56 (CD56) or cluster of differentiation 38(CD38) antigens are also highly expressed in multiple myeloma cells.With CD138 as the target for the treatment of CAR-T cells, several clinical studies have been registered, and the results show that some of them are effective.

In order to lay a foundation for the application of relapsed/refractory multiple myeloma patients with CAR-T therapy，objects are refractory/ relapsed patients with multiple myeloma,and plans to into the group of the number of cases in 50 cases.The main content is safety, efficacy and feasibility analysis of the CAR-T cells （single CAR-T or double CAR-T cells with BCMA、CD138、CD56 or CD38 ) in the treatment of refractory/relapsed multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

1. Relapsed/Refractory MM patients
2. Cell phenotype is BCMA/CD138/CD38/CD56 positive (single or combined) ,and minimal residual disease (MRD) was positive(cytology, genetic testing)
3. Estimated survival time is more than 3 months in multiple myeloma,and Karnofsky performance status(KPS) score is more than 60.
4. No cytapheresis and cell separation contraindication.
5. Hemoglobin is more than 80 gram per litre.
6. The function of important organ was satisfied:(1)cardiac ultrasound indicated that cardiac ejection fractions is more than 50%（EF≥50%）, and the electrocardiogram showed no obvious abnormality;(2)Blood oxygen saturation is more than 90%（SpO2≥90%）;(3)Creatinine（Cr） is less than 2.5 times normal range;(4)Alanine transaminase（ALT） and glutamic-oxalacetic transaminase（AST）is less than 3 times normal range,and total bilirubin is less than 2 milligram per deciliter(TBil≤2.0mg/dL).
7. After discussion by the expert group, the patient's condition was analyzed and combined with the general physical condition of the patient, the benefit of participating in the clinical trial was greater than the risk.
8. Volunteered for this clinical trail and signed a consent form .

Exclusion Criteria:

1. Patients with high tumor burden or progression of disease need to control the progression of disease in order to decrease the tumor burden.
2. Patients with active infection and fever.
3. Patients' neutrophilic granulocyte has decreased more than 10 days,and is difficult to control after treatment.
4. Patients are infected with fungus,bacteria or virus,and are difficult to control after treatment.
5. Patients with infection of HIV or with actively infection of Hepatitis B Virus(HBV) or Hepatitis C Virus(HCV).
6. Pregnant or lactating women.
7. Patients with severe insufficient cardiac, pulmonary and hepatorenal functions.
8. Patients had been treated with cell therapy but was invalid.After analyzing the patient's condition , the expert group think that the patient doesn't fit to attend the therapy of CART.
9. The monoclonal antibodies of BCMA or CD38 are invalid for the patients who have used the drug.
10. Any situation may do harm to the subjects or interfere the results.
11. After allogeneic transplantation, patients are more than 3 degrees of acute Graft-Versus-Host disease(GVHD).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Adverse events that Are related to treatment | 2 years
  Determine the toxicity profile of the BCMA/CD138/CD38/CD56-targeted CAR-T cells with Common Toxicity Criteria for Adverse Effects (CTCAE) version 4.0

SECONDARY OUTCOMES:
Estimate 2 year overall survival(OS) after infusion of BCMA/CD138/CD38/CD56-CART and sequential treatment | 2 years
  To estimate 2 year overall survival(OS) after BCMA/CD138/CD38/CD56-CART infusion and sequential treatment with Relapsed/Refractory MM
Estimate 2 year relapse rate after infusion of BCMA/CD138/CD38/CD56-CART and sequential treatment | 2 years
  To estimate 2 year relapse rate after BCMA/CD138/CD38/CD56-CART infusion and sequential treatment with Relapsed/Refractory MM
Estimate 2 year progression free survival after infusion of BCMA/CD138/CD38/CD56-CART and sequential treatment | 2 years
  To estimate 2 year progression free survival after BCMA/CD138/CD38/CD56-CART infusion and sequential treatment with Relapsed/Refractory MM

CONTACTS AND LOCATIONS:
Overall Officials: Yanjie He, Principal Investigator — Zhujiang Hospital
Locations (1):
- Southern Medical University Zhujiang Hospital, Guangdong, Guangdong, China

IPD SHARING:
Plan to Share IPD: No